CLINICAL TRIAL: NCT02196506
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of the Safety and Efficacy of Fixed-dose Brexpiprazole (OPC-34712) as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder With and Without Anxious Distress
Brief Title: Study of the Safety and Efficacy of Fixed-dose Brexpiprazole (OPC-34712) as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder With and Without Anxious Distress
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-13-214
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders
Keywords: OPC-34712; brexpiprazole; Major Depressive Disorder; Adjunctive Treatment; Anxious Distress
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders | interventions — Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brexpiprazole + ADT (Experimental): Brexpiprazole + ADT
  Interventions: Drug: Brexpiprazole +ADT
- Placebo + ADT (Placebo Comparator): Placebo + ADT
  Interventions: Drug: Placebo + ADT

INTERVENTIONS:
Drug: Placebo + ADT — Placebo + ADT Placebo + FDA Approved Antidepressant (ADT)
  Arms: Placebo + ADT
Drug: Brexpiprazole +ADT — Brexpiprazole + ADT Tablet, Oral, 2mg brexpiprazole and FDA Approved Antidepressant (ADT)
  Arms: Brexpiprazole + ADT

SUMMARY:
The purpose of this study is to assess the tolerability, safety, and efficacy of brexpiprazole (2.0 mg/day) as adjunctive therapy in adult subjects with a diagnosis of MDD with and without anxious distress

DETAILED DESCRIPTION:
The introduction of atypical antipsychotics has created a renewed interest in adjunctive therapy for MDD, particularly for treatment-resistant MDD. Several atypical antipsychotics have been shown to enhance the response to ADT. This is a phase 3, multicenter, randomized, double-blind, placebo-controlled, fixed-dose trial designed to assess the safety and efficacy of brexpiprazole (2.0 mg/day) as adjunctive therapy to an assigned open-label ADT in depressed subjects with and without anxious distress.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects between 18-65 years of age, with diagnosis of major depressive disorder with or without anxious distress
* Current depressive episode must be at least 8 weeks in duration

Exclusion Criteria:

* Subjects with a history of Neuroleptic Malignant Syndrome or Serotonin Syndrome
* Subjects who report an inadequate response to more than 3 antidepressant treatments in the current episode
* Subjects with a current Axis I diagnosis of: Delirium, dementia, amnestic or other cognitive disorder, Schizophrenia, schizoaffective disorder, or other psychotic disorder, Bipolar I or II disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudette Brewer, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (47):
- United States (30):
  - Birmingham, Alabama
  - Beverly Hills, California
  - Denver, Colorado
  - Hialeah, Florida
  - Orlando, Florida
  - Alpharetta, Georgia
  - Smyrna, Georgia
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Rochester Hills, Michigan
  - Cherry Hill, New Jersey
  - Jamaica, New York
  - New York, New York
  - Staten Island, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Edmond, Oklahoma
  - Portland, Oregon
  - Salem, Oregon
  - Philadelphia, Pennsylvania
  - Lincoln, Rhode Island
  - Columbia, South Carolina
  - Memphis, Tennessee
  - Wichita Falls, Texas
  - Murray, Utah
  - Woodstock, Vermont
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Spokane, Washington
- Germany (8):
  - Achim
  - Berlin
  - Düsseldorf
  - Frankfurt
  - Freiburg im Breisgau
  - Oranienburg
  - Stralsund
  - Würzburg
- Hungary (2):
  - Budapest
  - Győr
- Poland (4):
  - Gdansk
  - Lubin
  - Sosnowiec
  - Warsaw
- Slovakia (3):
  - Bratislava
  - Kosice-Barca
  - Liptovský Mikuláš

REFERENCES:
- [Derived] Kapadia S, Zhang Z, Ardic F, Patel M, Thase ME, Papakostas GI. Adjunctive brexpiprazole in patients with major depressive disorder who show minimal or partial response to antidepressant treatment: post hoc analysis of randomized controlled trials. Int J Neuropsychopharmacol. 2025 Oct 1;28(10):pyaf074. doi: 10.1093/ijnp/pyaf074. PMID 41055581
- [Derived] Ardic F, Zhang Z, Hogan M. Effects of adjunctive brexpiprazole in patients with major depressive disorder and sleep disturbance: a post hoc analysis of three randomized trials. Front Psychiatry. 2025 Aug 7;16:1618176. doi: 10.3389/fpsyt.2025.1618176. eCollection 2025. PMID 40852147
- [Derived] Kapadia S, Zhang Z, Csoboth C, Patel M, Thase ME, Papakostas GI. Adjunctive brexpiprazole in patients with unresolved symptoms of depression on antidepressant treatment who are early in the disease course: post hoc analysis of randomized controlled trials. Int J Neuropsychopharmacol. 2025 Aug 1;28(8):pyaf050. doi: 10.1093/ijnp/pyaf050. PMID 40607746
- [Derived] McIntyre RS, Bubolic S, Zhang Z, MacKenzie EM, Therrien F, Miguelez M, Boucher M. Effects of Adjunctive Brexpiprazole on Individual Depressive Symptoms and Functioning in Patients With Major Depressive Disorder and Anxious Distress: Post Hoc Analysis of Three Placebo-Controlled Studies. J Clin Psychopharmacol. 2024 Mar-Apr 01;44(2):133-140. doi: 10.1097/JCP.0000000000001825. PMID 38421922
- [Derived] Newcomer JW, Meehan SR, Chen D, Brubaker M, Weiss C. Changes in Metabolic Parameters and Body Weight in Patients With Prediabetes Treated With Adjunctive Brexpiprazole for Major Depressive Disorder: Pooled Analysis of Short- and Long-Term Clinical Studies. J Clin Psychiatry. 2023 Aug 28;84(5):23m14786. doi: 10.4088/JCP.23m14786. PMID 37656180
- [Derived] McIntyre RS, Therrien F, Ismail Z, Meehan SR, Miguelez M, Larsen KG, Chen D, MacKenzie EM, Thase ME. Effects of adjunctive brexpiprazole on patient life engagement in major depressive disorder: Post hoc analysis of Inventory of Depressive Symptomatology Self-Report data. J Psychiatr Res. 2023 Jun;162:71-78. doi: 10.1016/j.jpsychires.2023.04.012. Epub 2023 Apr 12. PMID 37099968
- [Derived] Newcomer JW, Eriksson H, Zhang P, Meehan SR, Weiss C. Changes in Metabolic Parameters and Body Weight in Patients With Major Depressive Disorder Treated With Adjunctive Brexpiprazole: Pooled Analysis of Phase 3 Clinical Studies. J Clin Psychiatry. 2019 Oct 1;80(6):18m12680. doi: 10.4088/JCP.18m12680. PMID 31577867
- [Derived] Hobart M, Zhang P, Weiss C, Meehan SR, Eriksson H. Adjunctive Brexpiprazole and Functioning in Major Depressive Disorder: A Pooled Analysis of Six Randomized Studies Using the Sheehan Disability Scale. Int J Neuropsychopharmacol. 2019 Mar 1;22(3):173-179. doi: 10.1093/ijnp/pyy095. PMID 30508090
- [Derived] Hobart M, Skuban A, Zhang P, Augustine C, Brewer C, Hefting N, Sanchez R, McQuade RD. A Randomized, Placebo-Controlled Study of the Efficacy and Safety of Fixed-Dose Brexpiprazole 2 mg/d as Adjunctive Treatment of Adults With Major Depressive Disorder. J Clin Psychiatry. 2018 May 22;79(4):17m12058. doi: 10.4088/JCP.17m12058. PMID 29873953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 837 participants at 51 trial sites in the following 5 countries:Germany,Hungary,Poland,Slovakia,andUnited States (US).A total of 1144 participants with major depressive disorder were screened for the trial, 837 enrolled into Phase A,394 were randomized into Phase B and 322 continued treatment with placebo+ADT in Phase A+
Pre-assignment Details: Trial consisted of a screening phase and 3 phases. In phase A (8-week single-blind prospective treatment phase) and in phase A+ (Single-blind phase A Responder), there was single treatment group. In phase B (6-week double-blind randomization phase), there were 2 treatment groups. All Outcome Measures were assessed in phase B.
Groups:
- Phase A: All ADT (Antidepressant Therapy): Participants meeting entrance criteria who were experiencing a major depressive episode with a HAM-D17 Total Score of greater than or equal 18 at baseline were enrolled into an 8-week Single-blind Prospective Treatment Phase (Phase A). All participants received single-blind placebo plus an investigator determined, open-label, ADT. Once assigned to an ADT by the investigator, participants remained on the same ADT for the duration of the trial. At the Week 8 visit, the IWRS (Interactive web response system) determined based on scores entered by the investigator, whether a participant was a "Phase A Responder" or a "Phase A Inadequate Responder."
- Phase B: Brexpiprazole + ADT: Participants received brexpiprazole 2 mg and ADT orally once daily for 6 weeks.
- Phase B: Placebo + ADT: Participants received matching placebo and ADT orally once daily for 6 weeks.
- Phase A +: ALL ADT: Phase A+ included participants who met criteria for a response at the end of the prospective treatment phase (Week 8 visit of Phase A) and participants who were not suitable for randomization in Phase B per the judgment of the investigator or medical monitor. Treatment response in Phase A was determined at the Week 8 visit based on improvement or lack of improvement of the participant's depressive symptoms, which was confirmed by clinical criteria that prospectively defined response. Participant response was determined from clinical data that were entered into the IWRS at each visit. Participants in Phase A+ received single-blind placebo+ADT for an additional 6 weeks, for a total of 14 weeks, and attended visits at Weeks 11 and 14.
Period: Phase A
Arm/Group | Phase A: All ADT (Antidepressant Therapy) | Phase B: Brexpiprazole + ADT | Phase B: Placebo + ADT | Phase A +: ALL ADT
Started | 837 | 0 | 0 | 0
Completed | 716 | 0 | 0 | 0
Not Completed | 121 | 0 | 0 | 0
Not completed — Participant Met Withdrawal Criteria | 34 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 34 | 0 | 0 | 0
Not completed — Adverse Event | 22 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0 | 0
Not completed — Protocol deviation | 12 | 0 | 0 | 0
Not completed — Participant withdrawn by investigator | 10 | 0 | 0 | 0
Period: Phase B
Arm/Group | Phase A: All ADT (Antidepressant Therapy) | Phase B: Brexpiprazole + ADT | Phase B: Placebo + ADT | Phase A +: ALL ADT
Started | 0 | 192 | 202 | 0
Completed | 0 | 177 | 196 | 0
Not Completed | 0 | 15 | 6 | 0
Not completed — Participant Met Withdrawal Criteria | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 2 | 0
Not completed — Withdrawal by Participant | 0 | 8 | 1 | 0
Not completed — Adverse Event | 0 | 4 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0
Period: Phase A+
Arm/Group | Phase A: All ADT (Antidepressant Therapy) | Phase B: Brexpiprazole + ADT | Phase B: Placebo + ADT | Phase A +: ALL ADT
Started | 0 | 0 | 0 | 322
Completed | 0 | 0 | 0 | 308
Not Completed | 0 | 0 | 0 | 14
Not completed — Participant Met Withdrawal Criteria | 0 | 0 | 0 | 1
Not completed — Withdrawal by Participant | 0 | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 6
Not completed — Participant withdrawn by investigator | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the participants from the Double-blind Randomization Phase
Groups:
- Brexpiprazole + ADT: Phase B: Brexpiprazole +Antidepressant therapy (ADT):
  Participants received brexpiprazole 2mg and ADT orally once daily for 6 weeks.
- Placebo + ADT: Phase B: Placebo + Antidepressant therapy (ADT):
  Participants received matching placebo and ADT orally once daily for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole + ADT | Placebo + ADT | Total
Number analyzed (Participants) | 192 | 202 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (12.7) | 42.7 (12.5) | 42.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 144 | 291
  Male | 45 | 58 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 181 | 192 | 373
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Hungary | 16 | 16 | 32
  United States | 100 | 106 | 206
  Poland | 26 | 26 | 52
  Slovakia | 23 | 25 | 48
  Germany | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in the Montgomery-Asberg Depression
Description: To assess the change in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score from Baseline (End of Phase A [Week 8]) to Week 14. The MADRS was utilized as the primary efficacy assessment of the participant's level of depression and was administered utilizing the Structured Interview Guide for the MADRS (SIGMA). The MADRS consisted of 10 items each with 7 defined grades of severity. The rater decided whether the rating lied on predefined scale steps (0, 2, 4, 6) or between them (1, 3, 5). The 10 items were apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The maximum total score was 60; 0, no symptom; 60, severely affected.
Time Frame: From baseline (end of Phase A [Week 8]) to week 14
Population: The primary analysis was performed on Efficacy Sample which included all randomized participants who took at least one dose of trial medication in Phase B and who have both an end of Phase A (Week 8) and at least one post-randomization MADRS Total Score during Phase B.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 191 | 202
Units on a scale | -10.4 (0.63) | -8.07 (0.61)
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Placebo + ADT; Statistical Analysis at Week 14; Test type: Superiority; p = 0.0074, Mixed Models Analysis; Mean Difference (Final Values) = -2.30, 95% CI 2-sided [-3.97 to -0.62]

2. Secondary Outcome: Change in the Sheehan Disability Scale (SDS) From Baseline to End of Treatment
Description: To assess the change in the Sheehan Disability Scale (SDS) Score (the mean of 3 individual item scores) from Baseline (End of Phase A [Week 8]) to Week 14 (End of Phase B). SDS was a 3-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life, and family life/home responsibility. Each item was scored using a scale of 0 to 10 (a higher score indicates symptoms have disrupted work, social life, and family life/home responsibility extremely). The maximum total score was 30; 0 = not at all, to 30 = extremely.
Time Frame: From baseline (end of Phase A [Week 8]) to week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 187 | 200
Units on a scale | -1.63 (0.18) | -1.41 (0.17)
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Placebo + ADT; Statistical Analysis at Week 14; Test type: Superiority; p = 0.3331, Mixed Models Analysis; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.66 to 0.23]

3. Secondary Outcome: Change From End of Phase A to End of Phase B in MADRS Total Score for the Subpopulation With <25% Improvement From Baseline of Phase A to End of Phase A in MADRS Total Score
Description: To assess the change from end of Phase A (Week 8 visit) to end of Phase B (Week 14 visit) in MADRS Total Score for the subpopulation with < 25% improvement from baseline of Phase A (Week 0) to end of Phase A (Week 8) in MADRS Total Score. The MADRS was utilized as the primary efficacy assessment of the participant's level of depression and was administered utilizing the Structured Interview Guide for the MADRS (SIGMA). The MADRS consisted of 10 items each with 7 defined grades of severity. The 10 items were apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The maximum total score was 60; 0, no symptom; 60, severely affected.
Time Frame: From baseline (end of Phase A [Week 8]) to week 14
Population: Subpopulation of <25% Improvement Sample: Comprised of all participants in the Efficacy Sample who had <25% improvement at the end of Phase A in MADRS Total Score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 161 | 158
Units on a scale | -11.1 (0.71) | -8.87 (0.71)
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Placebo + ADT; Statistical Analysis at Week 14; Test type: Superiority; p = 0.0263, Mixed Models Analysis; Mean Difference (Final Values) = -2.25, 95% CI 2-sided [-4.23 to -0.27]

4. Secondary Outcome: Change From End of Phase A to End of Phase B in MADRS Total Score for the Subpopulations With Anxious Distress as Specified in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V).
Description: To assess the change from end of Phase A (Week 8) to end of Phase B (Week 14) in MADRS Total Score for the subpopulations with anxious distress as specified in DSM-V. The MADRS was utilized as the primary efficacy assessment of the participant's level of depression and was administered utilizing the Structured Interview Guide for the MADRS (SIGMA). The MADRS consisted of 10 items each with 7 defined grades of severity. The 10 items were apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The maximum total score was 60; 0, no symptom; 60, severely affected.
Time Frame: From baseline (end of Phase A [Week 8]) to week 14
Population: Subpopulation of Anxious Distress Sample: Comprised of all participants in the Efficacy Sample who had anxious distress as specified in DSM-V.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 124 | 124
Units on a scale | -11.8 (0.81) | -8.87 (0.81)
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Placebo + ADT; Statistical Analysis at Week 14; Test type: Superiority; p = 0.0099, Mixed Models Analysis; Mean Difference (Final Values) = -2.98, 95% CI 2-sided [-5.24 to -0.72]

ADVERSE EVENTS:
Time Frame: Participants were assessed for the occurrence of adverse events (AEs) once the participant signed informed consent form through completion of the trial; up to 14-weeks after the participant entered the trial and actively monitored up to 30 (+2) days after their last dose of investigational medicinal product (this could be up to 22 weeks depending on duration of trial participation).
Description: Safety sample comprised of randomized participants in Phase B who received at least one dose of double-blind trial medication. No adverse events were assessed or collected from Phase A or A+ participants as those phases are single-blind, non-randomized, monotherapy treatment periods of the study and are outside of the pre-specified definition of the safety sample per the trial design.
Arm/Group | Brexpiprazole + ADT | Placebo + ADT
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/202
Serious Adverse Events (participants affected / at risk) | 1/192 | 0/202
Other Adverse Events (participants affected / at risk) | 49/192 | 35/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brexpiprazole + ADT (N=192) | Placebo + ADT (N=202)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brexpiprazole + ADT (N=192) | Placebo + ADT (N=202)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (11) | 10 (11)
Weight Increased (Investigations) | 10 (10) | 1 (1)
Akathisia (Nervous system disorders) | 16 (17) | 10 (12)
Headache (Nervous system disorders) | 7 (7) | 15 (24)
Restlessness (Psychiatric disorders) | 16 (16) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.